CLINICAL TRIAL: NCT03704246
Title: A Multicenter, Open and Phase II Clinical Study of HX008 for the Treatment in Patients With Advanced Solid Tumors
Brief Title: Recombinant Human Anti-PD-1 Monoclonal Antibody HX008 Injection for the Treatment of Advanced Solid Tumors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taizhou Hanzhong biomedical co. LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX008-II-02
Record Dates: First submitted 2018-10-07; First posted 2018-10-12 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-PD-1 (Other): Anti-PD-1 monoclonal antibody HX008 injection with a dose of 200mg (intravenous infusion, every 3 weeks)
  Interventions: Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Drug: Anti-PD-1 monoclonal antibody — HX008 is a monoclonal antibody drug which is intravenous drip at a dose of 200mg.
  Other Names: HX008

SUMMARY:
In this study, patients of advanced gastric adenocarcinoma with failed first-line chemotherapy-line or advanced mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) advanced solid carcinoma will be treated with HX008 combined with irinotecan and HX008 monotherapy There will be two cohorts in this study: Cohort 1 and Cohort 2. For Cohort 1, advanced gastric adenocarcinoma with failed first-line chemotherapy-line cancer participants, who had failed or were unable to tolerate first line chemotherapy with platinum-based or fluorouracil regimens. For Cohort 2, advanced solid tumor participants, who are required to have been previously treated with at least one line of systemic standard of care therapy.

DETAILED DESCRIPTION:
Cohort 1:

Currently, no PD-1 antibody against gastric cancer have been approved in China, and there are many patients with gastric cancer in China, so effective, low-toxicity and affordable treatment is urgently needed. This study aims to investigate the efficacy of combined application of recombinant human anti-PD-1 monoclonal antibody (HX008) and irinotecan in patients with locally advanced or metastatic gastric cancer (including gastric esophageal junction cancer) ,thus providing a better treatment for Chinese patients with gastric cancer.Advanced gastric adenocarcinoma with failed first-line chemotherapy-line cancer participants, who had failed or were unable to tolerate first line chemotherapy with platinum-based or fluorouracil regimens are needed.

Cohort 2:

Later-line therapies after failure of standard treatments for advanced solid cancer patients are limited. Mismatch repair (MMR) deficiency or microsatellite instability-high (MSI-H) played a role of positive predictive factor, which had been documented after the pembrolizumab and nivolumab trial were reported, for PD-1 blockade monotherapy in patients with advanced solid carcinomas.

In this study, patients with previously-treated locally-advanced or metastatic mismatched repair deficient (dMMR) or microsatellite instability-high (MSI-H) advanced solid tumors will be treated with HX008 monotherapy.Advanced solid tumor participants, who are required to have been previously treated with at least one line of systemic standard of care therapy are needed.

ELIGIBILITY:
Main inclusion Criteria:

1. Subject is male or female; ≥ 18 and ≤ 75 years of age for cohort 1 and ≥ 18 years of age for cohort 2 on the day of signing informed consent, and subject has voluntarily agreed to participate by giving written informed consent.
2. Subjects must have a histopathological diagnosis of any locally advanced or metastatic solid tumor, Subjects must have failed established standard medical anti-cancer therapies ( have disease progression after the therapies or be intolerant to the therapies) or Subjects refuse to standard therapies, or no effective treatment.
3. Subject must have a performance status of 0 to 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
4. Measurable disease as defined by RECIST v1.1.
5. Life expectancy ≥ 12 weeks.
6. Subject must have adequate hematologic and organ function.
7. Asymptomatic patients with Central Nervous System (CNS) metastasis or asymptomatic brain metastasis after treatment shall undergo computed tomography (CT) or magnetic resonance imaging (MRI) for no disease progression, stable for at least 3 months and no steroid treatment for at least 4 weeks.
8. Male subjects and female subjects should agree to take effective contraception from the date of signing the informed consent form until 3 months after the last administration.

Special inclusion criteria 1 in the Cohort 1.

1. Locally advanced or metastatic gastric adenocarcinoma (including gastric esophageal junction cancer) diagnosed histologically or cytologically.
2. Participants who had previously received a platinum-based or fluorouracil based first-line chemotherapy failed or could not tolerate.
3. The final cytotoxic drug, radiotherapy, or surgery≥4 weeks away. Special inclusion criteria 1 in the Cohort 2

1.Advanced malignant solid tumors confirmed by histology or cytology and confirmed as msi-h or dMMR by the central laboratory designated by the sponsor.

2.Participants must have received or not tolerated a first-line anti-tumor drug regimen.

Main exclusion Criteria:

1. Participants with other malignant tumors within 5 years before enrollment, excluding cured cervical carcinoma in situ and cured basal cell carcinoma of the skin.
2. Subject Is currently participating and receiving study therapy or has participated in a study of an investigational agent and receive study therapy within 28 days of the first dose of study drug.
3. Subject has not recovered to CTCAE Grade 1 or better from the adverse events due to cancer therapeutics administered.
4. Subject who had received anti-PD-1, PD-L1-,CTLA-4 monoclonal therapy, etc.
5. Subjects with active, or pre-existing, autoimmune diseases that may recur.
6. Systemic corticosteroids should be administered within 14 days before initial administration or during the study.
7. Subjects with active gastrointestinal ulcer, incomplete intestinal obstruction, active gastrointestinal hemorrhage and perforation.
8. Subjects with existing interstitial lung or pneumonia, pulmonary fibrosis, acute pulmonary disease, radioactive pneumonia;
9. Subjects with Uncontrollable and stable systemic diseases, such as cardiovascular and cerebrovascular diseases, diabetes, hypertension and tuberculosis.
10. Subjects with a history of infection with human immunodeficiency virus, or have other acquired or congenital immune deficiency diseases, or have a history of organ transplantation or stem cell transplantation.
11. Subject is positive for Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies), active hepatitis B (HBV surface antigen positive and HBV DNA ≥ 500 copies/ml)or hepatitis C or tuberculosis (HCV antibody positive).
12. Subjects with severe infection within 4 weeks before first administration, or those with active infection within 2 weeks before administration or intravenous antibiotic treatment.
13. Subjects who have been previously known to have severe allergic reactions to macromolecules/monoclonal antibodies or to any of the test drug components (CTCAE ≥Grade 3).
14. Participated in clinical trials of other drugs within 4 weeks before the first administration (subject to the use of the tested drugs).
15. Subjects with alcohol dependence or a history of drug abuse or drug abuse within one year.
16. Subjects with a clear history of neurological or mental disorders, such as epilepsy, dementia, poor compliance, or peripheral nervous system disorders;
17. Subjects with symptomatic brain metastases.
18. Women who are pregnant or lactating.
19. Subjects were not fit for other reasons concluded by the researchers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2018-09-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
ORR of HX008 combined with irinotecan and HX008 single drug | Up to approximately 2 years
  ORR was assessed according to Response Evaluation Criteria in Solid Tumors v 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
HX008 safety and tolerability assessed by monitoring AEs | From screening to up to 1 months after the last dose of study drug (up to approximately 2 years)
  Percentage of participants with adverse events (AEs), serious adverse events and AEs of special interest
Disease Control Rate (DCR) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vendor and investigator
Duration of Response (DOR) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vendor and investigator
Progression-Free Survival (PFS) | Up to approximately 2 years
  per RECIST 1.1 assessed by central imaging vedor and investigator
Overall Survival (OS) | Up to approximately 2 years
  Calculated by the Kaplan-Meier method.
Immunogenicity | From the first dose of study drug (up to approximately 2 years)
  Measured by MSD electroluminescence detection method

CONTACTS AND LOCATIONS:
Locations (30):
- China (30):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Yuhe Combination of Chinese Traditional and Western Medicine Recovery Hospital, Beijing
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu
  - Hunan Cancer Hospital, Changsha
  - Xiangya Hospital, Central South University, Changsha
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi
  - Fujian Cancer Hospital, Fuzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The affiliated Cancer Hospital of Harbin Medical University, Harbin
  - Anhui Provincial Cancer Hospital, Hefei
  - Shandong Cancer Hospital, Jinan
  - Jiangsu Provincial People's Hospital, Nanjing
  - Guangxi Medical University Cancer Hospital, Nanning
  - Fudan University Cancer Center, Shanghai
  - Liaoning Cancer Hospital, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Peking university shenzhen hospital, Shenzhen
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Cancer Hospital, Taiyuan
  - Tianjin Cancer Hospital, Tianjin
  - Tianjin People's Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - Wuhan Central Hospital, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xinxiang Medical College, Xinxiang
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang B, Song Y, Luo S, Yin X, Li E, Wang H, He Y, Liu Z, Fan Q, Liang X, Shu Y, Liu Y, Xu N, Zhang S, Zhuang Z, Zhang J, Kou X, Wang F, Zhu X, Zeng S, Wang K, Zhong H, Li S, Bai Y, Yu J, Dou Y, Ma T, Liu Q, Huang J. Pucotenlimab in patients with advanced mismatch repair-deficient or microsatellite instability-high solid tumors: A multicenter phase 2 study. Cell Rep Med. 2023 Dec 19;4(12):101301. doi: 10.1016/j.xcrm.2023.101301. Epub 2023 Nov 27. PMID 38016482
- [Derived] Song Y, Li N, Li Q, Liang X, Zhang S, Fan Q, Yin X, Zhuang Z, Liu Y, Zhang J, Kou X, Zhong H, Wang X, Dou Y, Huang J. HX008, an anti-PD1 antibody, plus irinotecan as second-line treatment for advanced gastric or gastroesophageal junction cancer: a multicenter, single-arm phase II trial. J Immunother Cancer. 2020 Oct;8(2):e001279. doi: 10.1136/jitc-2020-001279. PMID 33060149